CLINICAL TRIAL: NCT02465944
Title: A Phase II, Double-blind, Randomised, Placebo-controlled, Parallel Group Pilot Study to Evaluate the Safety and Efficacy of FFP104 in the Treatment of Subjects With Moderate to Severely Active Crohn's Disease
Brief Title: A Pilot Study of FFP104 in Subjects With Crohn's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fast Forward Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FFP104-002; 2015-001678-17 (EudraCT Number)
Record Dates: First submitted 2015-05-18; First posted 2015-06-09 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Crohn's Disease
Keywords: inflammation
MeSH Terms: conditions — Crohn Disease; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FFP104 - 2.5 mg/kg (Experimental): FFP104
  Interventions: Drug: FFP104
- FFP104 - 5.0 mg/kg (Experimental): FFP104
  Interventions: Drug: FFP104
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FFP104 — Three intravenous infusions of FFP104 over 15 days (d0, d7 and d14)
  Arms: FFP104 - 2.5 mg/kg; FFP104 - 5.0 mg/kg
Drug: Placebo — Three intravenous infusions of 0.9% Saline over 15 days (d0, d7 and d14)
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the safety, tolerability and efficacy of intravenously administered FFP104 or placebo over 15 days (3 total doses) in subjects with moderate to severely active Crohn's Disease

ELIGIBILITY:
Inclusion criteria

Subjects will be entered into this study only if they meet all of the following criteria:

* Willing and able to provide written informed consent.
* Willing and able to comply with all study procedures and visits.
* Male or female aged between 18 and 75 years, inclusive.
* Body Mass Index (BMI) between 18-35 kg/m2.
* Clinical diagnosis of Crohn's disease involving the colon and/or ileum for at least 3 months from Screening confirmed by radiological, endoscopic or histological evidence.
* Active Crohn's disease defined as a Crohn's Disease Activity Index (CDAI) score from 220 and 450, inclusive, at Screening.
* Active inflammatory disease as defined by Crohn's Disease Endoscopic Index of Severity (CDEIS) ≥ 8 (as determined by a Central Blinded Reader) at Screening.
* Tumor Necrosis Factor (TNF)-naïve or previously exposed to a single anti-TNF agent (such as infliximab, adalimumab or certolizumab pegol) with treatment discontinued at least 8 weeks prior to Screening due to inadequate response, loss of response or intolerance as judged by the Investigator.
* Must have adequate renal and hepatic function as adjudged by the Investigator.
* In good health (other than Crohn's disease) as evidenced by medical history and physical examination.

Exclusion criteria

Subjects will be entered into this study only if they meet none of the following criteria:

* Subjects who are pregnant, breastfeeding, or of child-bearing potential and not using a medically accepted form of contraception.
* Presence of fistulas, ileostomies, colostomies or rectal pouches or history of proctocolectomy or total colectomy. Subject has an ostomy or ileoanal pouch (subjects with a previous ileorectal anastomosis are not excluded).
* Subject has short bowel syndrome as determined by the Investigator.
* History of evidence of colonic mucosal dysplasia.
* Subject currently has a significant mechanical obstruction (stenosis).
* Subject has a current diagnosis of ulcerative or indeterminate colitis.
* Immunization with a live vaccine within 4 weeks of Screening, with the exception of influenza vaccine and no planned immunizations within the period of the study.
* Active or latent tuberculosis (TB) or tuberculosis infection; TB assessment and prophylaxis will be performed as per local biologicals regulations and guidelines.
* Subjects with a history of or ongoing chronic or recurrent infectious disease within the 12 months prior to Screening.
* Positive stool culture for Clostridium within the last 6 months prior to Screening.
* Use of prohibited medications/procedures, including;

  * Concomitant corticosteroids doses exceeding 20 mg/day of prednisone (equivalent)
  * Concomitant use of budesonide
  * Concomitant use of anti-TNF therapy
  * Subjects who received previous treatment with more than one anti-TNF agent
  * Concomitant use of cyclosporine, tacrolimus, sirolimus or mycophenolate mofetil
  * Prior or concomitant use of anti-α4 integrin or other non-TNF blocking biological
  * Use of tube or enteral feeding, elemental diet, or parenteral alimentation started within 2 weeks prior to Screening
  * Leukocytapheresis or granulocytapheresis within 2 weeks prior to Screening
* Use of any prescription medications/products (with the exception of prescription medications for contraception and/or medications deemed acceptable by the Investigator and Sponsor).
* Use of any over the counter (OTC), non-prescription preparations (including vitamins, minerals, phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to the Check-in visit (Day 0), unless deemed acceptable by the Investigator and Sponsor.
* Current or recent history (within 6 months of screening) of drug or substance abuse, including alcohol ≥ 14 units per week or who have a significant history of alcoholism or drug/chemical abuse within 6 months prior to the Screening visit (one unit of alcohol equals 0.5 pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1 shot [25 mL] of spirits).
* Subjects with known clinically significant cardiac disease (e.g., myocardial infarction or stroke within 6 months prior to Screening, unstable angina, claudication, etc.), or evidence of a clinically significant electrocardiogram (ECG) abnormality at Screening.
* A history of significant neurologic, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary or metabolic disease within 30 days of the Screening visit, as judged by the Investigator.
* Have a family history (more than one first degree relative) of multiple thrombotic events or a personal history of any venous or arterial thrombotic event including deep vein thrombosis, stroke, myocardial infarction, pulmonary embolus, and peripheral arterial thromboembolic events.
* Subject has had a positive hepatitis panel (including hepatitis B surface antigen [HBsAg], hepatitis B core antibody, and hepatitis C virus antibody [anti-HCV]) or a positive HIV antibody screen at time of Screening.
* Evidence of hepatic dysfunction, viral hepatitis, or current or chronic history of liver disease including non-alcoholic steatohepatitis (NASH) or abnormal hepatic markers (AST, ALT, ALP, or total bilirubin > 1.5 x upper limit of normal) at the time of the Screening visit.
* Abnormal renal function (BUN or creatinine >1.25 x upper limit of normal) at the time of the Screening visit.
* White Blood Cells <4 x 103/mm3; platelets <150 x 103/mm, hemoglobin < 6.2 mmol/L at the time of the Screening visit.
* Subjects with evidence of other serious, significant, acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.
* History of malignancy, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ.
* Active acute infection requiring systemic treatment for more than 2 weeks.
* Planned surgery during the study period or have undergone major surgery within the 3 months prior to the Screening visit.
* Subjects who have received any investigational drug within 60 days or use of other experimental anti-CD therapies within the last 30 days prior to Screening visit.
* Known sensitivity to any component of the study drug or previous sensitivity reaction or other clinically significant reaction to intravenous medications or biologic therapy.
* Subjects who have previously received FFP104 or have been previously enrolled in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed through clinical laboratory tests, vital signs, physical exams, and adverse event assessments | Up to 84 days

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical response (decrease of Crohn's Disease Activity Index (CDAI) score by ≥100 points from baseline) | Days 0, 7, 14, 28, 42 and 84
Proportion of subjects achieving clinical remission (attainment of absolute CDAI score of 150 points or less from baseline) | Days 0, 7, 14, 28, 42 and 84
Proportion of subjects achieving partial response (decrease of CDAI score by >70 points from baseline) | Days 0, 7, 14, 28, 42 and 84
Difference in CDAI score between FFP104 treated subjects and placebo subjects in each arm of the study | Days 0, 7, 14, 28, 42 and 84
Time to response (decrease in CDAI score by >100 points) | Days 0, 7, 14, 28, 42 and 84
Time to partial response (decrease of CDAI score by >70 points) | Days 0, 7, 14, 28, 42 and 84
Change from baseline in Crohn's Disease Endoscopic Index of Severity (CDEIS) | Day 42
Change from baseline in gut tissue organisation (histology) | Day 42
Percent change from baseline in faecal calprotectin level | Day 42
Percent change from baseline in C-Reactive Protein (CRP) levels | Day 7, 14, 28, 42 and 84
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | Day 42
Change from baseline in health outcome measures | Day 42
  Health outcome measures that will be used are Short Form 36 (SF36), the EuroQol EQ-5D-5L and the Work Productivity and Activity Impairment Questionnaire Crohn's Disease (WPAI-CD)
To evaluate changes from baseline in serum FFP104 levels | up to 84 days
To evaluate changes in lymphocyte sub-populations in peripheral blood | Day 0, 14 and 42

CONTACTS AND LOCATIONS:
Locations (2):
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Erasmus Medical Center, Rotterdam, Netherlands